CLINICAL TRIAL: NCT04956731
Title: Pharmacist Provision of Medication Abortion Pilot
Brief Title: Pharmacist Provision of Medication Abortion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Sarah Averbach, MD MAS, Associate Professor, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 210175
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-05

CONDITIONS: Abortion in First Trimester
Keywords: medication abortion, no-test medication abortion, pharmacist

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pharmacist provision of medication abortion (Experimental): This is a single arm study with 10 participants undergoing start to finish medication abortion provided by a pharmacist.
  Interventions: Other: Pharmacist Provision of Medication Abortion

INTERVENTIONS:
Other: Pharmacist Provision of Medication Abortion — Pharmacists providing start to finish medication abortions

SUMMARY:
This will be a pilot study among two pharmacists providing start to finish medication abortions to 10 patients utilizing a previously created toolkit. Following completion of the pilot, we will perform in-depth semi-structured interviews with the participating patients and pharmacists to understand their experiences with pharmacist provision of medication abortion. In addition, we will elicit feedback about ways to refine the toolkit to support the scale-up of pharmacist provision of medication abortion in the future.

DETAILED DESCRIPTION:
We will conduct a 'proof of concept' pilot study. Participating patients will be counseled by a trained pharmacist who will provide Mifepristone 200 mg and two doses of 800 mcg of Misoprostol. Patients will be instructed to take the 800 mcg of misoprostol buccally 24-48 hours after their Mifepristone. Patients whose estimated gestational age is between 64 and 70 days will be instructed to take the additional dose of 800 mcg of misoprostol 4 hours after the first dose. Patients who estimated gestational age is 63 days or less will be instructed to take the additional dose of 800 mcg of misoprostol if they do not experience at least moderate bleeding within the first 24 hours following their first misoprostol dose.

The standard Mifepristone consent form will be signed at this time and the patient will then be instructed to take the Mifepristone orally.

Participants will be contacted one week after receiving treatment by the providing pharmacist. If the participant history suggests concern for a continuing pregnancy, ectopic pregnancy or worrisome bleeding, they will be scheduled for in person evaluation. If the participant does not indicate any concern, they will be instructed to use the high sensitivity urine pregnancy test four weeks after taking their misoprostol. If the participant's first high sensitivity urine pregnancy test is positive but they have no symptoms concerning for ongoing pregnancy, they will be instructed to perform a second, high sensitivity urine pregnancy test in one week. If the second, high sensitivity urine pregnancy test is also positive, the patient will be evaluated in person.

We will continue our study by performing in-depth semi-structured interviews with the participating patients and pharmacists to understand their experiences and elicit feedback about ways to refine the toolkit. We will follow a prepared interview guide.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Pregnancy must be confirmed by either patient report of a positive urine pregnancy test, serum pregnancy test or ultrasound
* Patient's last menstrual period (LMP) must be less than 70 days before the anticipated date of mifepristone administration
* Patient must be certain of their LMP within 7 days and have regular menses
* Patient has no symptoms or risk factors for ectopic pregnancy including bleeding or spotting in the week before their visit, prior ectopic pregnancy, significant pelvic pain the last week, prior permanent contraception or tubal surgery, current intrauterine device (IUD) in place or IUD in place at time of conception.

Exclusion Criteria:

* Any contraindications to medication abortion, as reported on their medical history. These contraindicated include:

  1. Hemorrhagic bleeding disorder
  2. Current anticoagulation therapy
  3. Chronic adrenal failure
  4. Long-term systemic corticosteroid therapy
  5. Inherited porphyria

  d) Allergy to misoprostol or mifepristone
* Any patient with complex medical conditions will also be excluded from this initial pilot. These medical conditions include:

  1. Poorly controlled hypertension as defined a history of systolic blood pressure >160 or diastolic blood pressure >110 or patients requiring two or more antihypertensive medication to control their blood pressure. This will be exclusion criteria for the study but it not a standard exclusion criteria for medication abortion
  2. Poorly controlled diabetes as defined by a known history of Type 1 or Type 2 diabetes with history of finger stick blood sugar >200 or HbA1c>10 in the last 6 months. This will be exclusion criteria for the study but it not a standard exclusion criteria for medication abortion
  3. Hepatic or renal failure
  4. History of solid organ transplant
  5. 4 or more cesarean sections
  6. Allergy to NSAIDs.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Averbach, MD, MAS, Principal Investigator — UC San Diego Health
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sandoval S, Rafie S, Kully G, Mody S, Averbach S. Pharmacist provision of medication abortion: A pilot study. Contraception. 2024 Mar;131:110346. doi: 10.1016/j.contraception.2023.110346. Epub 2023 Dec 7. PMID 38065286
- See also: Pharmacist provision of medication abortion: A pilot study — https://doi.org/10.1016/j.contraception.2023.110346

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pharmacist Provision of Medication Abortion
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Pharmacist Provision of Medication Abortion
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — not recorded
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 0
    More than one race | 0
    Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Completion of Medication Abortion
Description: Negative Pregnancy Test
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacist Provision of Medication Abortion
Number analyzed (Participants) | 10
Participants | 9

2. Secondary Outcome: Patient Satisfaction, # of Patients Reporting "Very Satisfied"
Description: qualitative analysis of post abortion in depth interviews
Time Frame: 2 weeks following completion of medication abortion
Population: only 9 of the 10 participants completed post-abortion interview
Measure: Count of Participants; unit: Participants
Arm/Group | Pharmacist Provision of Medication Abortion
Number analyzed (Participants) | 9
Participants | 9

3. Secondary Outcome: Pharmacist Experience
Description: qualitative analysis of post pilot in depth interviews
Time Frame: 2 weeks following completion of all 10 medication abortion visits
Reporting Status: Not Posted

4. Secondary Outcome: Toolkit Changes
Description: per recommendation by participating pharmacists at post pilot in depth interviews
Time Frame: 2 weeks following completion of all 10 medication abortion visits
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Pharmacist Provision of Medication Abortion
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT04956731/Prot_SAP_000.pdf